CLINICAL TRIAL: NCT02462460
Title: Pilot Study Pancreatic and Ovarian Screening MR Imaging of Rapid With Motion Corrected T1, T2, and Advanced Diffusion Weighted Imaging for Patients With BRCA Mutation Who Undergo Screening Breast MRI
Brief Title: Rapid Pancreatic and Ovarian Screening MR Imaging With Motion Corrected T1, T2, and Advanced Diffusion Weighted Imaging for Patients With BRCA Mutation Who Undergo Screening Breast MRI
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-120
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Screening Breast MRI in Patients Who Are BRCA Mutation Carriers
Keywords: Breast MRI; T1 weighted and diffusion weighted MR; screening pancreatic; screening ovarian; 15-120

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with BRCA mutation: The purpose of this study is to optimize rapid pancreatic and ovarian MR screening protocols using T1, T2 and DW imaging sequences in BRCA mutation carriers. Each screening MR protocol is considered optimized if we reach 5 consecutive patients with technically adequate image quality. We will enroll up to 60 patients to perform the MR screening protocol, if the initial MR sequence parameters do not yield technically adequate MR images in a single patient, we will stop and modify our imaging protocol. We will continue to modify the technique until we reach 5 consecutive patients with technically adequate MR images for both on all imaging sequences. Thus, it is possible we will optimize different imaging sequences at different time points in our study. We plan to enroll at least 5 patients, and up to 60 patients with BRCA mutation who undergo breast MRI for this study. Participants will receive a copy of the questionnaire on the day of their Breast MRI.
  Interventions: Device: MRI; Behavioral: Optional Screening Questionnaire

INTERVENTIONS:
Device: MRI
Behavioral: Optional Screening Questionnaire

SUMMARY:
The purpose of this study is to create a rapid scan of the pancreas and ovaries that could be used in the future to screen patients at risk for pancreatic or ovarian cancers. Currently, Magnetic Resonance Imaging (MRI) examinations of the pancreas and ovaries can last 30-45 minutes each. The investigators hope to create a rapid pancreatic and ovarian MRI evaluation that can be used as a screening tool that is completed in approximately 15 minutes. They will compare different tools available on modern MRI scanners to see which one reliably offers high quality images of the pancreas and ovaries.

ELIGIBILITY:
A minimum of 5 and maximum of 60 evaluable patients will be imaged on this study. Description of the subject inclusion and exclusion criteria are listed below.

Inclusion Criteria:

* BRCA 1 or 2 mutation
* Age ≥ 30
* Patients scheduled to undergo screening breast MRI with contrast

Exclusion Criteria:

* Patients with known breast cancer
* Patients unable to complete their scheduled breast MRI
* Patients with prior pancreatic surgery or cancers
* Patients with prior ovarian cancer or surgery involving removal of one or both ovaries
* Patients with prior abdominal or pelvic surgery

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
define optimized acquisition | 1 year
  The images will be evaluated qualitatively for image quality from 1 to 5 with 5 = not adequate and 1 = adequate image quality by two radiologists in consensus. If both radiologists give a score of 1, the sequence will be considered to be adequate in image quality. Quantitative measurements of SNR will be performed on the pancreatic head, body and tail, and ovarian tissue by region of interest (ROI) analysis. Final acquisition times and spatial resolution for each sequence will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sawan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/